CLINICAL TRIAL: NCT02060435
Title: The Impact of the Epstein-Barr Virus Status on Clinical Outcome in Diffuse Large B Cell Lymphoma
Brief Title: Epstein-Barr Virus Status in Diffuse Large B Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, Professor, Samsung Medical Center
Other Study IDs: 2013-07-101-001
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: diffuse large B-cell lymphoma; Ebstein-Barr Virus
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — EBV RNA was detected by an in situ hybridization (ISH) technique using the EBV ISH kit (Leica Microsystems, Bannockburn, IL, USA).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- EBER+ AMC: EBV+DLBCL patients in Asan Medical Center
  Interventions: Other: EBER
- EBER+ SMC: EBV+DLBCL patients in Samsung Medical Center
  Interventions: Other: EBER
- EBER- SMC: EBV-DLBCL patients in Samsung Medical Center

INTERVENTIONS:
Other: EBER — EBV RNA was detected by an in situ hybridization (ISH) technique using the EBV ISH kit (Leica Microsystems, Bannockburn, IL, USA).
  Groups: EBER+ AMC; EBER+ SMC

SUMMARY:
The investigators analyzed clinical outcome in DLBCL patients according to age group to define the impact of EBV status on the clinical outcome.

DETAILED DESCRIPTION:
Epstein-Barr virus (EBV) positive diffuse large B-cell lymphoma (DLBCL) has been recognized as a new provisional entity in the 2008 World Health Organization (WHO) classification of tumors of hematopoietic and lymphoid tissue. This lymphoma is defined as EBV+ clonal B-cell proliferation in immunocompetent adults older than 50 years. To denote patient age in definition of this disease, age cutoff was defined as older than 50 years. However, this cutoff is clearly arbitrary without any scientific background. the knowledge on EBV+DLBCL in young adult is very scanty. This EBV+DLBCL in young adult can be the same disease entity or it can be a distinct disease form EBV+DLBCL of elderly.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed de novo DLBCL, according to the World Health Organization (WHO) classification:

  * registered in Samsung Medical Center (SMC) Lymphoma Cohort Study I/II (ClinicalTrials.gov Identifier: NCT00822731, NCT01877109) or identified from Asan Medical Center (AMC) medical database:
  * adequate amount and quality of paraffin-embedded biopsy specimen or unstained slides for EBV-encoded RNA (EBER) in situ hybridization.

Exclusion Criteria:

* Patients with unknown EBV status, primary central nervous system (CNS) lymphoma, post-transplant lymphoproliferative disorders (PTLDs), and HIV-positive DLBCL were excluded in the study.

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: (1) pathologically confirmed de novo DLBCL, according to the World Health Organization (WHO) classification: (ii) registered in Samsung Medical Center (SMC) Lymphoma Cohort Study I/II (ClinicalTrials.gov Identifier: NCT00822731, NCT01877109) or identified from Asan Medical Center (AMC) medical database: (iii) adequate amount and quality of paraffin-embedded biopsy specimen or unstained slides for EBV-encoded RNA (EBER) in situ hybridization.
Sampling Method: Probability Sample
Enrollment: 571 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
overall survival | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, MD PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Hong JY, Yoon DH, Suh C, Huh J, Do IG, Sohn I, Jo J, Jung SH, Hong ME, Yoon H, Ko YH, Kim SJ, Kim WS. EBV-positive diffuse large B-cell lymphoma in young adults: is this a distinct disease entity? Ann Oncol. 2015 Mar;26(3):548-55. doi: 10.1093/annonc/mdu556. Epub 2014 Dec 4. PMID 25475080